CLINICAL TRIAL: NCT00716040
Title: Effectiveness of a Social-Psychological Intervention to Improve Adherence to Antiretroviral Drug Regimens for AIDS: a Randomized Controlled Trial
Brief Title: Social-Psychological Intervention to Improve Adherence to HAART
Acronym: SPIAH-Q
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Maria Ines Battistella Nemes, Faculdade de Medicina da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2006-61277-6
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: AIDS; HIV Infections
Keywords: AIDS treatment; HAART adherence; intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will be submitted to four social-psychological individual sessions with a pre-trained health professional.
  Interventions: Behavioral: Social-psycho intervention to improve adherence to HAART
- Control (Other): The control group will be submitted to the usual care of the health service.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Social-psycho intervention to improve adherence to HAART — The intervention focus on the notion of scenes and scenarios to examine and discussing the experience of taking ARV medicines. In principle, such an approach provides a tool for conscientization, action and the invention of novel group and individual repertoires that may result in individual mobilization for improving adherence to treatment and reducing his/her vulnerability.
  Arms: Intervention
Other: Usual care — The control group will be submitted to the usual care of the health service
  Arms: Control

SUMMARY:
All eligible patients will be invited to use electronic monitoring of medication (MEMS) during the next six months. After two months with MEMS the enrolled patients will be randomized to intervention group or to control group. The intervention group will be submitted to four social-psycho sessions with a pre-trained health professional. The control group will receive the usual care of the health service.

The study will compare the rate of adherence to antiretroviral therapy between the intervention group and the control group. The duration of the study will be of six months. The analysis will be based on "intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old, with detectable viral load and more than six months under HAART

Exclusion Criteria:

* Pregnant women
* Patients participating in other trials
* Patients in treatment for hepatitis and for active opportunistic infection
* Patients with mental or physical condition which do not allow their attendance to the health service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Adherence to HAART | 24 weeks

SECONDARY OUTCOMES:
Viral Load | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ines B Nemes, PhD, Principal Investigator — Faculty of Medicine -University of Sao Paulo; Ernani T Santa Helena, PhD, Study Director — Regional University of Blumenau
Locations (1):
- Centro de Referência e Treinamento DST/AIDS, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Basso CR, Helena ET, Caraciolo JM, Paiva V, Nemes MI. Exploring ART intake scenes in a human rights-based intervention to improve adherence: a randomized controlled trial. AIDS Behav. 2013 Jan;17(1):181-92. doi: 10.1007/s10461-012-0175-4. PMID 22527264